CLINICAL TRIAL: NCT00333645
Title: Prophylaxis With Caspofungin for the Prevention of Invasive Fungal Infections in High-Risk Liver Transplant Recipients
Brief Title: Prophylaxis With Caspofungin in High-Risk Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Estudio de Infecciones en Transplantados (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GESITRA-01; 03-0409 (Spanish Drug Agency)
Record Dates: First submitted 2006-06-04; First posted 2006-06-06 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2006-12

CONDITIONS: Liver Transplantation; Fungal Infection
Keywords: Liver transplantation; Invasive fungal infection; Invasive aspergillosis; Prophylaxis; Caspofungin
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections | interventions — Caspofungin

INTERVENTIONS:
Drug: Caspofungin

SUMMARY:
This is a non-comparative, open, multisite prospective estimation study to evaluate the efficacy and safety of caspofungin in the prophylactic treatment of adults who have received an orthotopic liver transplant and are at high risk of developing an invasive fungal infection. It is expected that the proportion of high-risk liver transplant recipients who develop a documented (proven or probable per European Organization for Research and Treatment of Cancer/Mycoses Study Group [EORTC/MSG] modified criteria) invasive fungal infection during the first 100 days after the onset of prophylaxis with caspofungin will be lower than 15%. It is also expected that the incidence of serious drug-related adverse events will be less than 25%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient has received an orthotopic liver transplantation
* Patient meets criteria, as defined per protocol, for being considered at high risk of developing an invasive fungal infection post-liver transplantation
* For women of childbearing potential, patient must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Any systemic antifungal therapy (other than fluconazole for a maximum of 7 days) within 14 days of the administration of the study drug.
* Documented (proven/probable) or suspected (possible) invasive fungal infection at the time of enrollment.
* Abnormal laboratory values as defined per protocol.
* Allergy, hypersensitivity, or any serious reaction to an echinocandin antifungal.
* Patient not expected to survive at least 5 days.
* Patient is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-10; Study Completion 2007-03

PRIMARY OUTCOMES:
Absence of breakthrough proven/probable invasive fungal infection by day +100

SECONDARY OUTCOMES:
Absence of breakthrough proven/probable invasive aspergillosis by day +100
Discontinuation of study therapy due to a drug-related adverse event
Incidence of drug-related serious adverse event(s)
Incidence of drug-related adverse event(s)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Fortun, MD, Study Director — Hospital Ramon y Cajal, Madrid, Spain
Locations (13):
- Spain (13):
  - Complejo Hospitalario Juan Canalejo, A Coruña
  - Hospital de Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Complejo Hospitalario Carlos Haya, Málaga
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Result] Fortun J, Muñoz P, Cisneros JM, et al. Antifungal prophylaxis with caspofungin in high-risk liver transplant recipients: a noncomparative, open-label prospective clinical trial. Clinical Microbiology & Infection 12 (suppl. 4): P684, 2006. [Abstract on an interim analysis performed on the first 15 patients enrolled in the study, presented as a poster at 2006 ECCMID meeting].